CLINICAL TRIAL: NCT05831345
Title: Intraoperative Methadone for the Prevention of Postoperative Pain: a Randomized, Double-blind Clinical Study in Orthopedic Surgery
Brief Title: Intraoperative Methadone for the Prevention of Postoperative Pain
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Tatiana Besse-Hammer, Head Physician of the Clinical Research Unit, Brugmann University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CHUB-Methadone
Record Dates: First submitted 2023-04-14; First posted 2023-04-26 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Orthopedic Surgery
MeSH Terms: interventions — Methadone; Sufentanil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- S Group (Active Comparator): Patients receiving sufentanil during induction of general anesthesia
  Interventions: Drug: Sufentanil Citrate
- M Group (Experimental): Patients receiving methadone during induction of general anesthesia
  Interventions: Drug: Methadone Hydrochloride

INTERVENTIONS:
Drug: Methadone Hydrochloride — Classic induction of anesthesia (opioid, hypnotic and curare) but the team is blinded to the opioid used (sufentanil or methadone), which is prepared in identical syringes by the pharmacy
  Arms: M Group
Drug: Sufentanil Citrate — Classic induction of anesthesia (opioid, hypnotic and curare) but the team is blinded to the opioid used (sufentanil or methadone), which is prepared in identical syringes by the pharmacy
  Arms: S Group

SUMMARY:
The pain felt after orthopedic surgery in the absence of adequate locoregional anesthesia is often insufficiently controlled, especially during the first 24 hours postoperatively.

Methadone, due to its long half-life, may provide better pain control after orthopedic surgery when associated locoregional anesthesia cannot be performed.

It may be impossible to perform loco-regional anesthesia in various contexts: patient refusal, pre-existing neurological impairment, infection at the injection site, coagulopathies, inability to cooperate, total language barrier, allergy to anesthetics, unavailability of equipment (ultrasound, etc.) or equipped room, lack of experience of nursing staff in performing the block and in the postoperative management of the patient.

Intraoperative administration of methadone in these settings may be superior to sufentanil for pain control during the 24 hours post orthopedic surgery, and the pain control provided by methadone does not appear to imply a higher likelihood of adverse events related to opioids.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years old
* ASA 1-3 status
* Elective partial or total hip and knee arthroplasty

Exclusion Criteria:

* Patient refusal
* Preoperative renal failure (serum creatinine > 2 mg/dL or 1.5-fold
* Increase in basal plasma creatinine or GFR < 90 ml/min/1.73m2)
* Significant hepatic dysfunction (PT <50% or increase in 3 times basal transaminases)
* Known heart failure
* Preoperative hemodynamic instability (preoperative use of inotropes or vasopressors)
* Known methadone or sufentanil allergy
* Preoperative opioid use or history of opioid abuse
* Pregnancy and breastfeeding.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-02-28 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Total morphine consumption | 72 hours
  Total morphine consumption
Standard visual analogue scale (VAS) | 24 hours
  Pain is assessed using a standard visual analogue scale (VAS) in 11 points (from 0 (no pain) to 10 (worst pain))

SECONDARY OUTCOMES:
Patient satisfaction | 72 hours
  Patient satisfaction is assessed by means of a questionnaire at the end of hospital stay

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No